CLINICAL TRIAL: NCT05096169
Title: Pharmacokinetic Evaluation of Serum Testosterone Concentrations After Administration of Clomiphene Citrate
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-10022773
Record Dates: First submitted 2021-10-18; First posted 2021-10-27 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Testosterone Deficiency
MeSH Terms: interventions — Clomiphene

STUDY DESIGN:
Intervention Model Description: Individuals will be divided into two groups. Group 1 will receive clomiphene citrate at a dose of 25mg daily and will take one-half of a 50mg tablet daily. Group 2 will receive clomiphene citrate at a dose of 50mg every other day and will take one 50mg tablet every other day.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clomiphene citrate 25 mg daily for 12 weeks (Experimental)
  Interventions: Drug: Clomiphene Citrate 25mg
- Clomiphene citrate 50 mg every other day for 12 weeks (Experimental)
  Interventions: Drug: Clomiphene Citrate 50mg

INTERVENTIONS:
Drug: Clomiphene Citrate 25mg — clomiphene citrate at a dose of 25mg daily
  Arms: Clomiphene citrate 25 mg daily for 12 weeks
Drug: Clomiphene Citrate 50mg — clomiphene citrate at a dose of 50mg every other day
  Arms: Clomiphene citrate 50 mg every other day for 12 weeks

SUMMARY:
This is a randomized, open-label trial examining two doses of clomiphene citrate in men with low serum testosterone concentrations (total testosterone (TT) < 300 ng/dl).

DETAILED DESCRIPTION:
This is a randomized, open-label trial examining two doses of clomiphene citrate in men with low serum testosterone concentrations (total testosterone (TT) < 300 ng/dl). The investigators will perform a pharmacokinetic analysis of serum hormone concentrations (TT, LH, FSH, estradiol) after medication administration. Researchers hypothesize that testosterone levels will increase in both groups and this may allow to dose clomiphene citrate so that patients do not need to take the medication daily.

ELIGIBILITY:
Inclusion Criteria:

* Male, 21-45 years of age
* Serum testosterone concentration < 300 ng/dl measured on two separate occasions (separated by at least one week), with collection prior to 10AM

Exclusion Criteria:

* Serum testosterone concentration > 300 ng/dl
* Abnormal serum prolactin (PRL) concentration (PRL > 15.2 ng/ml)
* Concurrent or prior use of hormone-modifying medications (clomiphene citrate or other SERM, testosterone replacement therapy or other testosterone-containing products/treatments, gonadotropin therapy, aromatase inhibitors, estrogen-containing products/treatments)
* Documented karyotype abnormality
* Diagnosis of Kallmann syndrome
* Any prior chemotherapy, radiation therapy to the groin/pelvis, or known exposure to gonadotoxic agents
* History of cryptorchidism or prior orchiopexy
* History of testicular cancer or prior orchiectomy
* History of pituitary tumor or resection of pituitary tumor
* History of prostate cancer or severe benign prostatic hypertrophy
* History of epididymitis or epididymo-orchitis, or orchitis (including mumps)
* History of primary hypogonadism
* History of prior urinary tract infection
* History of intravenous drug use
* Any of the following comorbidities: renal insufficiency, heart disease, peptic ulcer disease, cerebrovascular disease, liver disease, psychiatric disorders, chronic pain, bleeding diatheses, anemia, polycythemia, vision problems
* Medical history or concurrent illness that the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial, or constitutes an unacceptable risk to the subject
* Documented allergy or hypersensitivity to clomiphene citrate or other SERM

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum testosterone | Evaluation will occur at baseline, day 2, day 4, weeks 1 - 4, and again at weeks 8, 12, and 16.
  Change in serum testosterone

SECONDARY OUTCOMES:
Change in FSH levels | Evaluation will occur at baseline, day 2, day 4, weeks 1 - 4, and again at weeks 8, 12, and 16.
  Serum levels of follicle-stimulating hormone (FSH)
Change in LH levels | Evaluation will occur at baseline, day 2, day 4, weeks 1 - 4, and again at weeks 8, 12, and 16.
  Serum levels of luteinizing hormone (LH)
Change in estradiol levels | Evaluation will occur at baseline, day 2, day 4, weeks 1 - 4, and again at weeks 8, 12, and 16.
  Serum levels of estradiol levels

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulligan T, Frick MF, Zuraw QC, Stemhagen A, McWhirter C. Prevalence of hypogonadism in males aged at least 45 years: the HIM study. Int J Clin Pract. 2006 Jul;60(7):762-9. doi: 10.1111/j.1742-1241.2006.00992.x. PMID 16846397
- [Background] Mulhall JP, Trost LW, Brannigan RE, Kurtz EG, Redmon JB, Chiles KA, Lightner DJ, Miner MM, Murad MH, Nelson CJ, Platz EA, Ramanathan LV, Lewis RW. Evaluation and Management of Testosterone Deficiency: AUA Guideline. J Urol. 2018 Aug;200(2):423-432. doi: 10.1016/j.juro.2018.03.115. Epub 2018 Mar 28. PMID 29601923
- [Background] Wheeler KM, Sharma D, Kavoussi PK, Smith RP, Costabile R. Clomiphene Citrate for the Treatment of Hypogonadism. Sex Med Rev. 2019 Apr;7(2):272-276. doi: 10.1016/j.sxmr.2018.10.001. Epub 2018 Dec 3. PMID 30522888
- [Background] Mazzola CR, Katz DJ, Loghmanieh N, Nelson CJ, Mulhall JP. Predicting biochemical response to clomiphene citrate in men with hypogonadism. J Sex Med. 2014 Sep;11(9):2302-7. doi: 10.1111/jsm.12592. Epub 2014 Jun 5. PMID 24902614
- [Background] Moskovic DJ, Katz DJ, Akhavan A, Park K, Mulhall JP. Clomiphene citrate is safe and effective for long-term management of hypogonadism. BJU Int. 2012 Nov;110(10):1524-8. doi: 10.1111/j.1464-410X.2012.10968.x. Epub 2012 Mar 28. PMID 22458540
- [Background] Katz DJ, Nabulsi O, Tal R, Mulhall JP. Outcomes of clomiphene citrate treatment in young hypogonadal men. BJU Int. 2012 Aug;110(4):573-8. doi: 10.1111/j.1464-410X.2011.10702.x. Epub 2011 Nov 1. PMID 22044663
- [Background] Tenover JS, Bremner WJ. The effects of normal aging on the response of the pituitary-gonadal axis to chronic clomiphene administration in men. J Androl. 1991 Jul-Aug;12(4):258-63. PMID 1917692
- [Background] Bendre SV, Murray PJ, Basaria S. Clomiphene Citrate Effectively Increases Testosterone in Obese, Young, Hypogonadal Men. Reprod Syst Sex Disord. 2015 Dec;4(4):155. doi: 10.4172/2161-038X.1000155. Epub 2015 Nov 13. PMID 26844009
- [Background] Habous M, Giona S, Tealab A, Aziz M, Williamson B, Nassar M, Abdelrahman Z, Remeah A, Abdelkader M, Binsaleh S, Muir G. Clomiphene citrate and human chorionic gonadotropin are both effective in restoring testosterone in hypogonadism: a short-course randomized study. BJU Int. 2018 Nov;122(5):889-897. doi: 10.1111/bju.14401. Epub 2018 Jun 14. PMID 29772111
- [Background] Ramasamy R, Scovell JM, Kovac JR, Lipshultz LI. Testosterone supplementation versus clomiphene citrate for hypogonadism: an age matched comparison of satisfaction and efficacy. J Urol. 2014 Sep;192(3):875-9. doi: 10.1016/j.juro.2014.03.089. Epub 2014 Mar 21. PMID 24657837
- [Background] Krzastek SC, Sharma D, Abdullah N, Sultan M, Machen GL, Wenzel JL, Ells A, Chen X, Kavoussi M, Costabile RA, Smith RP, Kavoussi PK. Long-Term Safety and Efficacy of Clomiphene Citrate for the Treatment of Hypogonadism. J Urol. 2019 Nov;202(5):1029-1035. doi: 10.1097/JU.0000000000000396. Epub 2019 Oct 9. PMID 31216250
- [Background] Knight JC, Pandit AS, Rich AM, Trevisani GT, Rabinowitz T. Clomiphene-Associated Suicide Behavior in a Man Treated for Hypogonadism: Case Report and Review of The Literature. Psychosomatics. 2015 Sep-Oct;56(5):598-602. doi: 10.1016/j.psym.2015.06.003. Epub 2015 Jun 12. No abstract available. PMID 26362915
- [Background] Pasqualotto FF, Fonseca GP, Pasqualotto EB. Azoospermia after treatment with clomiphene citrate in patients with oligospermia. Fertil Steril. 2008 Nov;90(5):2014.e11-2. doi: 10.1016/j.fertnstert.2008.03.036. Epub 2008 Jun 16. PMID 18555230
- [Background] Ernst S, Hite G, Cantrell JS, Richardson A Jr, Benson HD. Stereochemistry of geometric isomers of clomiphene: a correction of the literature and a reexamination of structure-activity relationships. J Pharm Sci. 1976 Jan;65(1):148-50. doi: 10.1002/jps.2600650140. No abstract available. PMID 1255423
- [Background] Murdter TE, Kerb R, Turpeinen M, Schroth W, Ganchev B, Bohmer GM, Igel S, Schaeffeler E, Zanger U, Brauch H, Schwab M. Genetic polymorphism of cytochrome P450 2D6 determines oestrogen receptor activity of the major infertility drug clomiphene via its active metabolites. Hum Mol Genet. 2012 Mar 1;21(5):1145-54. doi: 10.1093/hmg/ddr543. Epub 2011 Nov 22. PMID 22108178
- [Background] Goldstein SR, Siddhanti S, Ciaccia AV, Plouffe L Jr. A pharmacological review of selective oestrogen receptor modulators. Hum Reprod Update. 2000 May-Jun;6(3):212-24. doi: 10.1093/humupd/6.3.212. PMID 10874566
- [Background] Ghobadi C, Mirhosseini N, Shiran MR, Moghadamnia A, Lennard MS, Ledger WL, Rostami-Hodjegan A. Single-dose pharmacokinetic study of clomiphene citrate isomers in anovular patients with polycystic ovary disease. J Clin Pharmacol. 2009 Feb;49(2):147-54. doi: 10.1177/0091270008328096. Epub 2008 Nov 25. PMID 19033451
- [Background] Mikkelson TJ, Kroboth PD, Cameron WJ, Dittert LW, Chungi V, Manberg PJ. Single-dose pharmacokinetics of clomiphene citrate in normal volunteers. Fertil Steril. 1986 Sep;46(3):392-6. doi: 10.1016/s0015-0282(16)49574-9. PMID 3091405
- [Background] Fontenot GK, Wiehle RD, Podolski JS. Differential effects of isomers of clomiphene citrate on reproductive tissues in male mice. BJU Int. 2016 Feb;117(2):344-50. doi: 10.1111/bju.13244. Epub 2015 Sep 7. PMID 26220499
- [Background] Adashi EY. Clomiphene citrate: the case for a monoisomeric preparation. Baillieres Clin Obstet Gynaecol. 1993 Jun;7(2):331-47. doi: 10.1016/s0950-3552(05)80134-8. No abstract available. PMID 8358894
- [Background] Wiehle R, Cunningham GR, Pitteloud N, Wike J, Hsu K, Fontenot GK, Rosner M, Dwyer A, Podolski J. Testosterone Restoration by Enclomiphene Citrate in Men with Secondary Hypogonadism: Pharmacodynamics and Pharmacokinetics. BJU Int. 2013 Jul 12;112(8):1188-200. doi: 10.1111/bju.12363. Online ahead of print. PMID 23875626
- [Background] Kim MJ, Byeon JY, Kim YH, Kim SH, Lee CM, Jung EH, Chae WK, Lee YJ, Jang CG, Lee SY, Choi CI. Effect of the CYP2D6*10 allele on the pharmacokinetics of clomiphene and its active metabolites. Arch Pharm Res. 2018 Mar;41(3):347-353. doi: 10.1007/s12272-018-1005-7. Epub 2018 Mar 7. PMID 29516347